CLINICAL TRIAL: NCT06466707
Title: Collectie Van Microbioomstalen Van Huid, Mond, Vagina en Feces Van Gezonde Westerse Donoren Voor Fundamenteel en Functioneel Microbioom-onderzoek.
Brief Title: Collection of Microbiome Samples of Healthy Western Donors for Fundamental and Functional Microbiome Research
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ONZ-2023-0659
Record Dates: First submitted 2024-05-21; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collection of microbiome samples (Other): Collection of skin, oral and vaginal (if applicable) microbiome samples by means of a swab and collection of fecal material using Fecotainer collection kit. No treatments will be given to the healthy volunteers.
  Interventions: Other: Collection of microbiome samples

INTERVENTIONS:
Other: Collection of microbiome samples — Collection of skin, oral and vaginal (if applicable) microbiome samples by means of a swab and collection of fecal material using Fecotainer collection kit.

SUMMARY:
Large numbers of micro-organisms (especially bacteria) live in and on human bodies and have a very important function for the health. These microorganisms are called 'the microbiota'. They aid in the digestion of food, ensure the production of certain vitamins, and are very important for the development and regulation of the immune system. In many diseases (including Crohn's disease, arthritis, obesity, diabetes and cancer), a disruption of microbial composition is observed. There are indications that a disruption of the microbiome can contribute to the development of inflammatory diseases and cancer, but the underlying processes are not sufficiently understood. To understand the mechanisms underlying these disease processes, fundamental research is conducted at Ghent University. Stool, skin, oral and vaginal samples from various origins are examined, e.g. from people from indigenous tribes with a traditional lifestyle. It is important that these samples can be compared with microbiome samples from healthy Western (West-European) controls. In this study, the investigators want to build up a collection of samples from healthy donors between the ages of 2 and 70, with the exception of vaginal samples collected from women between the ages of 18 and 45. The samples will form the basis for further fundamental and functional research into microbiota-host interactions at Ghent University.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Age between 2 and 70 years old
* Dutch speaking
* West-European origin

Exclusion Criteria:

* Diagnosis of chronic disease (such as osteoarthritis, rheumatoid arthritis, diabetes, Crohn's disease, inflammatory bowel disease (IBD), asthma, COPD, etc.)
* Antibiotics taken within 3 months before sampling

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Composition of the microbiome, as determined by metagenomics analysis of the skin, oral, vaginal and fecal microbiome samples | 4 years
  Characterization of skin, oral, vaginal and fecal microbiome profiles from Western donors versus indigenous Brazilian tribes (Yanomami, samples collected previously)
Compostition of the metabolome, as deteremined by metabolomics analysis skin, oral, vaginal and fecal microbiome samples | 4 years
  Characterization of skin, oral, vaginal and fecal metabolome profiles from Western donors versus indigenous Brazilian tribes (Yanomami, samples collected previously)
Measurement of disease progression upon administration of different microbiota (Western versus indigenous) by weight measurement | 4 years
  Measurement of disease progression in arthritis, colorectal cancer, intestinal inflammation, obesity, etc. by measuring weight loss or gain.
Measurement of disease progression upon administration of different microbiota (Western versus indigenous) by detecting blood in stool | 4 years
  Measurement of disease progression in colorectal cancer, intestinal inflammation, etc. by determining presence of blood in stool samples.
Measurement of disease progression upon administration of different microbiota (Western versus indigenous) by determining stool consistency | 4 years
  Measurement of disease progression in colorectal cancer, intestinal inflammation, etc. by determining stool consistency.
Measurement of disease progression upon administration of different microbiota (Western versus indigenous) by serum glucose measurement | 4 years
  Measurement of disease progression in obesity by measuring serum glucose concentrations.
Measurement of immune activation upon administration of different microbiota (Western versus indigenous). | 4 years
  Measurement of immune cell composition by means of flow cytometry analysis.
Identification of the micro-organisms from different microbiota (Western versus indigenous) linked to disease progression. | 4 years
  Identification of microorganisms involved in disease models (including arthritis, colorectal cancer, intestinal inflammation, obesity, etc.) by means of in-vitro and in-vivo models. The stool samples are administered to mouse models of various diseases via oral gavage, after which the disease process is closely studied. For the in-vitro models, these samples are used to stimulate cell lines to investigate the effect on, for example, T cell activation, macrophage polarization or general cell proliferation.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Verhasselt, MD-PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD will be collected in a pseudonymised database (spreadsheet), the link to the participant's identity is maintained separately from the study data. This pseudonymised data may be shared with other researchers, however, the link to the participan's identity will only be known by the PI and research team of Prof. Lars Vereecke.
Supporting Information: Study Protocol, CSR